CLINICAL TRIAL: NCT00887913
Title: Clinical Study to Evaluate the Performance of Fractional Radiofrequency for Improvement of Skin Texture Via Skin Resurfacing and Wrinkles Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Yehudit Kraizer, Syneron Medical
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Matrix RF_Facial Tx
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Results first posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Skin Resurfacing; Wrinkle Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Fractional RF treatment with Matrix RF applicator — 3 treatments, single pass, 2-50J
  Other Names: Matrix RF Applicator

SUMMARY:
The purpose of this study is to determine whether the Matrix RF applicator is effective in the treatment of facial skin texture and wrinkle reduction.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent agreement signed by the subject.
* Healthy males or females older than 21 years of age.
* Having at least two facial sub-areas with visible lines/wrinkles and elastosis, which correlate to a score of 2 6 on the Fitzpatrick Classification of Wrinkling and Degree of Elastosis.
* Fitzpatrick skin type I-VI (note: skin type VI should not undergo treatment using resurfacing procedure parameters).
* Willingness to follow the treatment and follow-ups schedule and the post-treatment care.
* For female candidates - post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study (i.e., oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide, or abstinence).

Exclusion Criteria:

* Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breastfeeding.
* Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
* Having a permanent implant in the treated area, such as metal plates and screws, or an injected chemical substance.
* Having a history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treated area, unless treatment is conducted following a prophylactic regimen.
* Having received acne treatment with a light-based device within 1 month of treatment or during the study.
* Use of isotretinoin (Accutane®) within 6 months of treatment or during the study.
* Use of non-steroidal anti-inflammatory drugs (NSAIDS, e.g., ibuprofen-containing agents) one week before and after each treatment session.
* Use of retinoids, antioxidants or skin nourishing supplements within 2 months of treatment or during the study.
* Having received a facial dermabrasion or chemical peel treatment within 3 months of treatment or during the study.
* Having received treatment with light, RF or other devices in the treated area within 6 months of treatment or during the study.
* Having received Botox/collagen/fat injections or other methods of augmentation with injected or implanted material in the treated area within 9 months of treatment or during the study.
* Having undergone a resurfacing procedure, face lift or eyelid surgery within a year of treatment or during the study.
* Having undergone any other surgery in the treated area within 6 months of treatment (or more if skin has not healed completely) or during the study.
* History of keloid scarring or of abnormal wound healing.
* Suffering from current or history of significant skin conditions in the treated area or inflammatory skin conditions, including, but not limited to: excessive skin dryness, psoriasis, eczema, rash, rosacea (particularly severe open wound stage), indurate acne, varicella scars, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course.
* History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
* History of epidermal or dermal disorders (particularly if involving collagen or microvascularity).
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
* Suffering from hormonal imbalance, as per the Investigator's discretion.
* Having a known anticoagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course (to allow inclusion, temporary cessation of use as per the subject's physician discretion).
* Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions.
* Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), or pertinent neurological disorders.
* Vascular lesion, tattoo or permanent make-up in the treated area.
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
* Participation in a study of another device or drug within one month prior to enrollment or during the study.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Advanced Dermatology, Lincolnshire, Illinois
  - Laser and Dermatology Surgery Center, Chesterfield, Missouri
- Laserderm, Ottawa, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Treatment group- undergo 3 treatments every 4-6 weeks
Period: Overall Study
Arm/Group | Treatment
Started | 69
Completed | 63
Not Completed | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 65
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 51.02 (8.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 45
  Canada | 24

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Fine Lines
Description: Improvement of fine lines (wrinkles) assessed per anatomical area treated based on Improvement Scale: 0-4 where higher scores indicate a better outcome.
  Improvement is graded by means of photographs taken at baseline vs treatment 3 and baseline vs 6week follow up
Time Frame: 4 week follow up after last treatment
Population: Per protocol each defined anatomical area treated was assessed for improvement according to Improvement Scale- 0-4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Fine Lines
Arm/Group | Treatment
Number analyzed (Participants) | 63
Number analyzed (Fine Lines) | 162
Scores on a scale | 1.77 (0.98)

2. Primary Outcome: Improvement in Smoothness
Description: Smoothness of anatomical treated area assessed based on Improvement Scale 0-4.Where higher scores indicate a better outcome.
  Improvement is graded by means of photographs taken at baseline vs treatment 3 and baseline vs 6week follow up
Time Frame: 4 weeks follow up post last treatment
Population: Analysis was per protocol, each area treated was graded on its improvement regarding the smoothness of the skin
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Smoothness
Arm/Group | Treatment
Number analyzed (Participants) | 63
Number analyzed (Smoothness) | 162
Scores on a scale | 1.90 (1.05)

3. Primary Outcome: Improvement in Brightness
Description: Assess the improvement in brightness of the treated anatomical area using Improvement Scale where higher scores indicate a better outcome.
  Improvement is graded by means of photographs taken at baseline vs treatment 3 and baseline vs 6week follow up
Time Frame: 4 week follow up post last treatment
Population: Per protocol, each anatomical area treated was assessed for skin brightness using the Improvement Scale of 0-4 where 0= 0%, 1= 1-25%, 2=26-50%, 3=51-75%, 4= 76-100% based on before and photographs. Maximum value grade is 4 and the minimum value grade is 0.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Brightness
Arm/Group | Treatment
Number analyzed (Participants) | 63
Number analyzed (Brightness) | 162
Scores on a scale | 1.68 (1.18)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the study, up to 5 months
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is under a general confidentiality agreement and must have prior written approval by the Sponsor prior to publishing the study results.